CLINICAL TRIAL: NCT02111954
Title: PET/CT Study of GRP Receptors With Ga-68-NODAGA-MJ9 in Prostate Cancer Compared to F-18-FCH PET / CT
Brief Title: Ga-68-NODAGA-MJ9 Compared to F-18-FCH PET/CT for Prostate Cancer Patients
Status: Completed | Type: Observational
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, John O. Prior, Nuclear Medicine Department, University of Lausanne Hospitals
Other Study IDs: 402/12
Record Dates: First submitted 2014-04-09; First posted 2014-04-11 (Estimated); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; primary; recurrence; F-18-FCH PET/CT; Ga-68-NODAGA-MJ9 PET/CT
MeSH Terms: conditions — Prostatic Neoplasms; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- F-18-FCH & Ga-68-NODAGA-MJ9: 1 PET/CT with F-18-FCH + 1 PET/CT with Ga-68-NODAGA-MJ9
  Interventions: Diagnostic Test: 1 PET/CT with F-18-FCH + 1 PET/CT with Ga-68-NODAGA-MJ9

INTERVENTIONS:
Diagnostic Test: 1 PET/CT with F-18-FCH + 1 PET/CT with Ga-68-NODAGA-MJ9 — Each patient will have two PET/CT
  Other Names: 1 PET/CT with F-18-FCH; 1 PET/CT with Ga-68-NODAGA-MJ9

SUMMARY:
Prostate cancer patients for whom a F-18-FCH PET/CT is indicated. Ga-68-NODAGA-MJ9 is a new PET/CT radiotracer aiming at giving complementary information : more precise images and early localisation of recurrence to standard imaging

DETAILED DESCRIPTION:
Patient with primary or relapsing prostate cancer for whom F-18-FCH PET/CT is indicated will be proposed to participate to the present study. After signing the patient informed consent, both F-18-FCH and Ga-68-NODAGA-MJ9 PET/CT will be scheduled with a maximum 10 day-interval.

No adverse events are expected.

ELIGIBILITY:
Inclusion Criteria:

* Age : adult patients
* Karnofsky : ≥ 80%
* Patients with histologically proven prostate cancer for whom 18F-fluocholine PET/CT is indicated for primary cancer staging, or for recurrence with increase of blood PSA. In order to provide a detection probability of 30% or more, a blood PSA 0.5 ng / ml or more in post initial curative intent surgery will be required.
* Signed informed consent.

Exclusion Criteria:

* Lack of discernment to sign the consent form
* Age <18 years
* Patient under hormonal treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with proven prostate cancer
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2014-04; Primary Completion 2016-10-28 (Actual); Study Completion 2016-10-28 (Actual)

PRIMARY OUTCOMES:
Positivity of the new radiotracer Ga-68-NODAGA-MJ9 compared to the standard radiotracer F-18-FCH | At baseline (after F-18-FCH PET/CT)
  PET images : SUVmax, SUVmean, VOI (mL), SUV41% lesions/ SUVbackground CT images : size lesions measured in 3D (axial, coronal and sagittal), density in Hounsfield Units (HU)

CONTACTS AND LOCATIONS:
Overall Officials: John O. Prior, MD, PhD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gnesin S, Cicone F, Mitsakis P, Van der Gucht A, Baechler S, Miralbell R, Garibotto V, Zilli T, Prior JO. First in-human radiation dosimetry of the gastrin-releasing peptide (GRP) receptor antagonist 68Ga-NODAGA-MJ9. EJNMMI Res. 2018 Dec 12;8(1):108. doi: 10.1186/s13550-018-0462-9. PMID 30543050